CLINICAL TRIAL: NCT06496581
Title: A Randomized Phase III Trial Evaluating the Efficacy and Safety of Standard of Care +/- 177Lu-PSMA617 in de Novo Metastatic Hormone-sensitive Prostate Cancer Patients Having a PSA≥0.2 ng/mL at 6-8 Months After Systemic Treatment Initiation
Brief Title: Standard of Care +/- 177Lu-PSMA-617 In de Novo mHSPC Patients With Poor PSA Response (PEACE6-Poor Responders)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GTG-2301 (GETUG-AFU 42); 2022-502408-57-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer Metastatic
Keywords: Genital Diseases, Male; Prostatic Diseases; Hormones; 177Lu-PSMA-617; PSA
MeSH Terms: conditions — Genital Diseases, Male; Prostatic Diseases | interventions — Pluvicto; Standard of Care; Androgen Antagonists; Prednisone; apalutamide; enzalutamide; Radiotherapy; Docetaxel; darolutamide

STUDY DESIGN:
Intervention Model Description: Phase III, international, multicenter, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Control arm): Standard of Care (SoC) alone (Active Comparator): The SoC is defined as one the following treatment which was initiated 6 to 8 months ahead of inclusion in this trial and still ongoing at the time of the randomization and continued at least until the CRPC stage is reached.:
  * ADT with an ARSI (i.e. abiraterone + prednisone, or apalutamide, or enzalutamide) ± radiotherapyª
  * ADT with docetaxelᵇ plus an ARSI (i.e. abiraterone + prednisone, or darolutamide,) ± radiotherapyª
  ª Radiotherapy can be part of any standard treatment aforementioned as long as it is not PSMA-based and completed at least 4 weeks ahead of randomization OR planned right after randomization in arm A.
  ᵇ Whenever docetaxel was part of the systemic treatment initiation, its administration must have been completed at least 4 weeks ahead of randomization.
  Interventions: Drug: Standard of Care
- Arm B (Experimental arm): 177Lu-PMSA-617 + SoC (Experimental): Once every 6 weeks, 7400 MBq 177Lu-PMSA-617 will be administered for up to a total of 4 cycles. Upon 177Lu-PMSA-617 treatment completion, the ongoing standard systemic treatment is to be maintained and continued at least until the CRPC stage is reached.
  The SoC is defined as one the following treatment which was initiated 6 to 8 months ahead of inclusion in this trial and still ongoing at the time of the randomization:
  * ADT with an ARSI (i.e. abiraterone + prednisone, or apalutamide, or enzalutamide) ± radiotherapyª
  * ADT with docetaxelᵇ plus an ARSI (i.e. abiraterone + prednisone, or darolutamide,) ± radiotherapyª
  ª Radiotherapy can be part of any standard treatment aforementioned as long as it is not PSMA-based completed at least 4 weeks ahead of randomization OR planned right after 177Lu-PSMA-617 in arm B.
  ᵇ Whenever docetaxel was part of the systemic treatment initiation, its administration must have been completed at least 4 weeks ahead of randomization.
  Interventions: Drug: 177Lu-PMSA-617; Drug: Standard of Care

INTERVENTIONS:
Drug: 177Lu-PMSA-617 — Once every 6 weeks, 7400 MBq 177Lu-PMSA-617 will be administered for up to a total of 4 cycles.
  Other Names: Pluvicto®
  Arms: Arm B (Experimental arm): 177Lu-PMSA-617 + SoC
Drug: Standard of Care — ADT, abiraterone and each ARSI (Apalutamide, Darolutamide, Enzalutamide) will be administrated according to the standard of care
  Other Names: ADT with an ARSI (i.e. abiraterone + prednisone, or apalutamide, or enzalutamide) ± radiotherapy* or ADT with docetaxel* plus an ARSI (i.e abiraterone + prednisone, or darolutamide,) ± radiotherapy

SUMMARY:
PEACE-6 Poor Responders is an international, multicenter, open-label, controlled, randomized, phase III trial to evaluate the efficacy and safety of 177Lu-PSMA-617 when administered on top of the ongoing standard systemic treatment compared to standard systemic treatment alone in patients with de novo metastatic hormone-sensitive prostate cancer (mHSPC) who do not present with a satisfactory response characterized by a serum prostatic specific antigen (PSA) level of ≥ 0.2 ng/mL at 6 to 8 months after systemic treatment initiation for mHSPC (i.e. poor responders) in the absence of evidence of cancer progression (including a rising PSA level).

DETAILED DESCRIPTION:
The study plans to enroll 500 patients over 63 months who will be randomized (1:1) to receive either: (i) Control arm: SoC (ADT+ ARSI (second-generation androgen receptor signaling inhibitors) +/- RT or ADT+ ARSI +/- RT) or (ii) Experimental arm: 177Lu-PSMA-617 + SoC (ADT+ ARSI +/- RT or ADT+ docetaxel + ARSI +/- RT). Response to treatment will be assessed according to the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria. Treatment will be continued at least until castration-resistant prostate cancer (CRPC) stage is reached, defined by evidence of cancer progression (either a confirmed PSA rise or a radiographic progression) with serum testosterone being at castrated levels (<0.50 ng/mL). This systemic treatment may be continued after CRPC is reached, based on patient benefit and the investigator's opinion. Treatment may also be terminated at the initiative of either the patient or the investigator for any reason that would be beneficial to the patient, including: unacceptable toxicity, intercurrent conditions that preclude continuation of treatment, or patient request. At the end of treatment period, the follow-up period will last for 102 months (8.5 years). The overall trial duration, including the follow-up, is expected to last 18.5 years.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met ahead of randomization to satisfy trial eligibility requirements:

1. Signed a written informed consent form prior to any trial specific procedures.

   Note: In case of physical incapacitation, a trusted representative of their choice, which is not the Investigator or sponsor, can sign on the behalf of the patients.
2. Aged ≥18 years old
3. Life expectancy > 6 months as per investigator estimate
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
5. Men with histologically or cytologically confirmed adenocarcinoma of the prostate
6. De novo metastatic disease defined by clinical or radiographic evidence of metastases at diagnosis (i.e. before any treatment started). If not available, a more recent imaging can be used
7. Measurable disease or bone lesions evaluable according to PCWG3 criteria. Patients with doubtful bone metastases are not eligible
8. A pre-randomization 68Ga-PSMA-11 PET/CT scan performed within 4 weeks prior to randomization in the trial.

   FDG PET scan is not required for this protocol. All patients will be treated independently from the results of pre-randomization PSMA PET scan: patients with PSMA-positive or PSMA-negative disease according to PROMISE 2.0 criteria are eligible.
9. Have 6 to 8 months of previous AND ongoing standard systemic treatment for prostate cancer consisting in either:

   * ADT with an androgen receptor signaling inhibitor (ARSI) (i.e., abiraterone (plus prednisone), or apalutamide or enzalutamide) ± radiotherapy **
   * ADT with docetaxel* plus an ARSI (i.e. abiraterone (plus prednisone), or darolutamide,) ± radiotherapy**

   Note:

   *Docetaxel must have been stopped at least 4 weeks ahead of randomization.

   ** Previous radiotherapy to the primary tumor and/or to the metastases is accepted as long as it was not PSMA-based and must has been completed at least 4 weeks ahead of randomization.
10. Stable or declining PSA level but not a rising one
11. Serum PSA of ≥ 0.2 ng/mL at 6 to 8 months after systemic treatment initiation
12. Testosterone level < 50 ng/dl or < 1.7 nmol/L
13. Be fit enough for 177Lu-vipivotide tetraxetan treatment:

    * Adequate bone marrow function: hemoglobin ≥90 g/L (in absence of red blood cell transfusion within 4 weeks prior to randomization), absolute neutrophil count ≥1.5 x10⁹/L, platelet count >100 x10⁹/L
    * Adequate liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.0 x upper limit of normal (ULN), or ≤ 5.0 x ULN in the presence of liver metastases; bilirubin <1.5 x ULN (unless known or suspected Gilbert syndrome, then <3 x ULN is permitted)
    * Adequate renal function: calculated creatinine clearance ≥ 50 ml/min (using the MDRD or CKD EPI method).
14. For sexually active men with female partners of reproductive potential or with pregnant women, agreement to use a condom with another effective contraceptive method during trial participation and up to 14 weeks after study treatment completion.
15. Affiliated to the social security system or in possession of equivalent private health insurance (according to local regulations for participation in clinical trials).
16. Willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up.

Exclusion Criteria:

Patients presenting with any of the following criteria are not eligible:

1. Any evidence of cancer progression (including a rising PSA level, clinical progression, or radiological progression)
2. Prior or concurrent PSMA-based radioligand therapy or other PSMA target treatments
3. Known hypersensitivity to the components of the study therapy or its analogs
4. Any condition preventing the use of the standard of care and/or specific experimental treatments tested in the trial
5. Any of the following within 6 months before randomization: stroke, myocardial infraction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure New York Heart Association (NYHA) Class III or IV
6. Hypertension not controlled by an anti-hypertensive treatment (systolic blood pressure [sBP] ≥ 160 mmHg or diastolic blood pressure [dBP] ≥ 95 mmHg, 3 consecutive measures taken 5 minutes apart)
7. Severe or uncontrolled concurrent disease, infection or co-morbidity
8. Pathological findings consistent with small cell carcinoma of the prostate
9. History of malignancy within 3 years of the current diagnosis with the exception of successfully treated basal cell or squamous cell skin carcinoma
10. Ongoing participation in another clinical trial involving an investigational product.. Treatment with an investigational product must have ended within 28 days prior to the day of randomization
11. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons
12. Persons deprived of their liberty or under protective custody or guardianship

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2033-02-01 (Estimated); Study Completion 2039-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death due to any cause, up to 8.5 years
  Overall survival (OS) is defined as the time from the date of randomization to the date of death due to any cause.
Radiographic progression-free survival (rPFS) | From randomization to radiographic progression or death, up to 8.5 years
  Radiographic progression-free survival (rPFS) is defined as the time from randomization to the date of radiographic progression according to PCWG3 criteria by investigator assessment, or death, whichever occurs first.

SECONDARY OUTCOMES:
Castration-Resistance Prostate Cancer-Free Survival (CRPC-FS) | From randomization to onset of castration-resistance or death, up to 8.5 years
  Castration-Resistance Prostate Cancer-Free Survival (CRPC-FS) is defined as the time from randomization to the onset of castration-resistance or death from any cause, whichever occurs first.
Prostate Cancer-Specific Survival (PCSS) | From the date of randomization to a PCSS event, up to 8.5 years
  Prostate Cancer-Specific Survival (PCSS) is defined as the time from the date of randomization to the date of death due to prostate cancer.
PSA response | From baseline over the treatment period, up to 8.5 years
  PSA response will be assessed by the maximum change of PSA (rise or fall) from baseline over the treatment period. A complete PSA response is defined by an undetectable level of serum PSA.
Skeletal-related event-free survival (SRE-FS) | From randomization to the onset of a SRE-FS event, up to 8.5 years
  Skeletal-related event-free survival (SRE-FS) is defined as the time from the randomization date to the date of diagnosis of either a skeletal-related event (SRE) (fracture, or bone pain requiring radiation therapy, or spinal cord compression, or preventive surgery to the bones) or death, whichever occurs first.
Time to severe urinary event (SUE) | From randomization to the onset of a SUE event, up to 8.5 years
  Time to severe urinary event (SUE) is defined as the time from the randomization date to the date of diagnosis of either one of the following SUE, whichever occurs first: urinary retention with need for a urinary catheter, suprapubic catheter, double J stent, nephrostomy, treatment of the prostate by radiotherapy or trans-urethral resection of the prostate (TURP) or prostatectomy done to relieve patients with local symptoms.
Time to initiation of first subsequent anti-cancer systemic therapy for CRPC (TTSST1) | From randomization to initiation of the first anti-cancer systemic therapy for CRPC, up to 10 years
  TTSST1 is defined as the time from the randomization date to the date of initiation of the first anti-cancer systemic therapy for CRPC.
Time to initiation of second subsequent anti-cancer systemic therapy for CRPC (TTSST2) | From randomization to initiation of the second anti-cancer systemic therapy for CRPC, up to 10 years
  TTSST2 is defined as the time from the randomization date to the date of initiation of the second anti-cancer systemic therapy for CRPC.
Efficacy of first subsequent anti-cancer systemic therapy for CRPC | From first anti-cancer systemic therapy for CRPC to disease progression or death, up to 10 years
  Efficacy of subsequent anti-cancer systemic therapy for CRPC will be defined as the time from first anti-cancer systemic therapy for CRPC to disease progression or death from any cause, whichever comes first.
Efficacy of second subsequent anti-cancer systemic therapy for CRPC | Fromsecond anti-cancer systemic therapy for CRPC to disease progression or death, up to 10 years
  Efficacy of second subsequent anti-cancer systemic therapy for CRPC will be defined as the time from second anti-cancer systemic therapy for CRPC to disease progression or death from any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, MD, Study Chair — Gustave Roussy, Villejuif; Gwenaelle GRAVIS, MD, Study Chair — IPC, Marseille
Locations (25):
- France (25):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Bergonié, Bordeaux
  - CHRU Brest, Brest
  - Centre Francois Baclesse, Caen
  - CHU Henri Mondor, Créteil
  - Centre Georges-François Leclerc, Dijon
  - CHU Grenoble, Grenoble
  - Centre Léon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHRU Nancy, Nancy
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - Hôpital Saint Louis, Paris
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Rouen, Rouen
  - Institut Curie, Saint-Cloud
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - ICANS, Strasbourg
  - IUCT Oncopole, Toulouse
  - CHRU Tours, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon request to the sponsor
Supporting Information: Study Protocol, CSR
Time Frame: After primary analysis until end of trial
Access Criteria: Steering committee approval